CLINICAL TRIAL: NCT04687501
Title: The Effect of Virtual Reality on Anxiety and Pain in Patients Undergoing Gynecological Surgery; a Randomised Controlled Trial
Brief Title: Effect of VR on Anxiety and Pain in Gynecological Surgery
Acronym: VRAP-G
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Principal Investigator, Ilse Bekkers, Drs, Zuyderland Medisch Centrum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL72290.096.20
Record Dates: First submitted 2020-03-03; First posted 2020-12-29 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Pain, Postoperative; Anxiety; Pain Catastrophizing; State Anxiety
Keywords: Postoperative pain; Anxiety; State anxiety; Pain catastrophizing; Analgesic use
MeSH Terms: conditions — Pain, Postoperative; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR-group (Experimental): The participants randomised into this group can choose for an immersive guided relaxation VR experience or an interactive VR experience. The VR intervention is additional to the standard postoperative care management, the standard pain protocol is explained below.
  The VR-intervention will be given using the Oculus Go Virtual Reality glasses with touchpad.
  Interventions: Device: Virtual Reality
- Standard care-group (No Intervention): The participants randomized into the standard care- group will receive the usual standard pre-and postoperative management.
  Standard pain protocol:
  1. Preoperative (arrival day-care unit) start with 1000mg paracetamol orally administered.
  2. Postoperative Meloxicam 15mg orally administered, or when oral medication is not possible (due to nausea e.g.) than diclofenac supp 100mg or diclofenac i.v. 75mg.
  3. On recovery ward, when necessary depending on pain score (NRS>4): dipidolor 2.5-5mg i.v. and 10-15mg i.m. after consulting the anesthesiologist.
  4. Postoperative at home 4dd1000mg paracetamol will be continued, in combination with meloxicam 1dd15mg during 3 days. Also tramadol 50mg with a maximum of 4dd will be prescribed.

INTERVENTIONS:
Device: Virtual Reality — Virtual reality in gynaecological surgery in the pre- and postoperative setting
  Arms: VR-group

SUMMARY:
Rationale: Lack of postoperative acute pain management is associated with increased morbidity, longer recovery time, more opioid use and subsequently increased health care costs. There is increasing evidence virtual reality (VR) is effective in the reduction of acute pain. Alternative methods to reduce postoperative pain and multimodal analgesia are necessary for acute postoperative pain management and to reduce opioid use and their adverse effects.

Objective: The aim of this study is to explore the effect of VR on pain in the immediate postoperative period after elective gynecological surgery.

Secondary objectives are evaluating pre-and postoperative anxiety, pain catastrophizing, analgesic use, length of hospital stay between both groups and to explore tolerability, feasibility and satisfaction of VR use.

Study design: The study concerns a non-blinded, single centre, randomised controlled trial.

Study population: Eligible women fulfill the inclusion criteria and receive elective gynecological surgery in the Zuyderland Medical Centre location Heerlen.

Intervention: The study population will be randomly divided into the intervention group (VR-group) or the standard care- group. The intervention group can choose for an immersive guided relaxation VR experience or an interactive VR experience during the pre- and postoperative period additional to the usual standard care. The participants randomised to the standard care- group will receive only the usual standard care pre-and postoperative.

Main study parameters: The primary outcome is postoperative pain measured on a numeric rating scale (NRS). A total of 30 patients have to be included in each group. This means that a total of 60 women will have to be included in the study.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

The study population experiences a small medical risk when participating to this study. They can experience side-effects of VR for example dizziness or nausea and in rare cases epileptic insults.

Participants of the study have to fill in a questionnaire before randomization and pre-and postoperative score of pain and anxiety on a zero to ten score scale.

DETAILED DESCRIPTION:
"An unpleasant sensory and emotional experience associated with actual or potential tissue damage, or described in terms of such damage", this is the definition of pain according to the International Association for the Study of Pain (IASP). Severe post-operative pain is experienced by approximately 50-80% of the patients.

Lack of postoperative acute pain management is associated with increased morbidity, longer recovery time, more opioid use and subsequently increased health care costs. Postoperative pain can cause a higher morbidity, because of cardiovascular, pulmonic and gastro-intestinal problems.

Besides, surgery and acute pain are both independent risk factors for the development of chronic pain. The reduction of acute pain and therefore managing postoperative pain may contribute to the prevention of chronic pain.

In general, nowadays, medication is the treatment of choice for acute pain and mainly opioid analgesics are used for pain relief. Worldwide this contributes to excessive drug dependence and opioid abuse. Opioid use comes with several negative side effects, for example a potential delay in recovery and an increased risk of permanent disability.

Nowadays, new methods related to pain management are developed. For example, Virtual reality (VR) is an upcoming technology used within healthcare. It is thought that the perception of pain is related to the amount of attention that is given to pain stimuli. The theory behind the working mechanism of VR to reduce pain is that VR acts as a distraction to limit the user's processing of nociceptive stimuli, by stimulating the visual cortex in the brain. In 2000, Hoffman published the first preliminary evidence for the beneficial effect of VR in reducing pain in a burn care unit. They also showed a trend to experience less anxiety during VR use. In the next upcoming years, a growing body of research was done to explore the effects of VR.

A recent systematic review and meta-analysis showed VR to be an effective treatment for reducing acute pain. Next to being effective in reducing pain, it is also a proven useful tool in reducing preoperative anxiety. VR can be used as a safe, non-invasive, analgesic method, without risks of drug addiction and minimum side effects.

In this study, the investigators want to explore the effect of VR on postoperative pain in patients undergoing elective gynecological surgery as a serious alternative for pain medication. The investigators hypothesize VR will reduce post-operative pain and consequently postoperative opioid use and anxiety reduction.

ELIGIBILITY:
Inclusion Criteria:

* Written and orally given informed consent
* 18 years and older
* Native Dutch speaker
* Indication for elective gynecological surgery under spinal anesthesia
* No contra-indication to anesthesia:

Exclusion Criteria:

* Chronic pain patients; defined as 'persistent or recurrent pain lasting longer than 3 months' . The pain is not due to the gynecological problem.
* Chronical use of pain medication (opioids)
* History of prior opioid use defined as use within 8 to 90 days prior to the surgical procedure
* Alcohol or drug abuse
* Known car sickness
* Epileptic insults in previous history
* Psychotically seizures in previous history
* Claustrophobic
* Blindness
* History of mental illness

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-09 (Actual)

PRIMARY OUTCOMES:
NRS pain | immediately after surgery
  reduction in postoperative pain score (NRS, numeric rating scale). Scaling from 0-10, where 0 means no pain and 10 means the worst imaginable pain

SECONDARY OUTCOMES:
STAI (State-Trait Anxiety Inventory) questionnaire (6 questions) | baseline
  Pre-operative anxiety. The score ranges from 20 to 90 and the higher the score the more anxiety the person experiences
Pain Catastrophizing Scale questionnaire | baseline
  Pain catastrophizing. The subscales of the PCS can be calculated separately or overall with a maximum total score of 52. The higher the score, the more catastrophizing thoughts are present.
NRS anxiety | baseline and immediately after surgery
  Difference in anxiety scores pre-and post VR intervention. Scaling on a scale form 0 to 10, where 0 means no anxiety and 10 means the worst imaginable anxiety
Analgesic use | Within 24-48hours after surgery
  daily use of paracetamol, NSAIDs, opioids
Length of hospital stay | within 24-48hours after surgery
  Length of hospital stay
VR Questionnaire | within 24hours after surgery
  Tolerability, feasibility and satisfaction of VR use
NRS pain preoperative | baseline
  Preoperative pain score (NRS). Scaling from 0-10, where 0 means no pain and 10 means the worst imaginable pain

CONTACTS AND LOCATIONS:
Overall Officials: Martine Wassen, Dr, Principal Investigator — Zuyderland Medical Centre
Locations (1):
- Zuyderland Medical Centre, Heerlen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Treede RD. The International Association for the Study of Pain definition of pain: as valid in 2018 as in 1979, but in need of regularly updated footnotes. Pain Rep. 2018 Mar 5;3(2):e643. doi: 10.1097/PR9.0000000000000643. eCollection 2018 Mar. PMID 29756089
- [Background] Popping DM, Zahn PK, Van Aken HK, Dasch B, Boche R, Pogatzki-Zahn EM. Effectiveness and safety of postoperative pain management: a survey of 18 925 consecutive patients between 1998 and 2006 (2nd revision): a database analysis of prospectively raised data. Br J Anaesth. 2008 Dec;101(6):832-40. doi: 10.1093/bja/aen300. Epub 2008 Oct 22. PMID 18945716
- [Background] Gan TJ. Poorly controlled postoperative pain: prevalence, consequences, and prevention. J Pain Res. 2017 Sep 25;10:2287-2298. doi: 10.2147/JPR.S144066. eCollection 2017. PMID 29026331
- [Background] Joshi GP, Ogunnaike BO. Consequences of inadequate postoperative pain relief and chronic persistent postoperative pain. Anesthesiol Clin North Am. 2005 Mar;23(1):21-36. doi: 10.1016/j.atc.2004.11.013. PMID 15763409
- [Background] Mills SEE, Nicolson KP, Smith BH. Chronic pain: a review of its epidemiology and associated factors in population-based studies. Br J Anaesth. 2019 Aug;123(2):e273-e283. doi: 10.1016/j.bja.2019.03.023. Epub 2019 May 10. PMID 31079836
- [Background] Zhao S, Chen F, Feng A, Han W, Zhang Y. Risk Factors and Prevention Strategies for Postoperative Opioid Abuse. Pain Res Manag. 2019 Jul 10;2019:7490801. doi: 10.1155/2019/7490801. eCollection 2019. PMID 31360271
- [Background] Mallari B, Spaeth EK, Goh H, Boyd BS. Virtual reality as an analgesic for acute and chronic pain in adults: a systematic review and meta-analysis. J Pain Res. 2019 Jul 3;12:2053-2085. doi: 10.2147/JPR.S200498. eCollection 2019. PMID 31308733
- [Background] Spiegel B, Fuller G, Lopez M, Dupuy T, Noah B, Howard A, Albert M, Tashjian V, Lam R, Ahn J, Dailey F, Rosen BT, Vrahas M, Little M, Garlich J, Dzubur E, IsHak W, Danovitch I. Virtual reality for management of pain in hospitalized patients: A randomized comparative effectiveness trial. PLoS One. 2019 Aug 14;14(8):e0219115. doi: 10.1371/journal.pone.0219115. eCollection 2019. PMID 31412029
- [Background] Hoffman HG, Patterson DR, Carrougher GJ. Use of virtual reality for adjunctive treatment of adult burn pain during physical therapy: a controlled study. Clin J Pain. 2000 Sep;16(3):244-50. doi: 10.1097/00002508-200009000-00010. PMID 11014398
- [Background] Dehghan F, Jalali R, Bashiri H. The effect of virtual reality technology on preoperative anxiety in children: a Solomon four-group randomized clinical trial. Perioper Med (Lond). 2019 Jun 4;8:5. doi: 10.1186/s13741-019-0116-0. eCollection 2019. PMID 31171963
- [Background] JahaniShoorab N, Ebrahimzadeh Zagami S, Nahvi A, Mazluom SR, Golmakani N, Talebi M, Pabarja F. The Effect of Virtual Reality on Pain in Primiparity Women during Episiotomy Repair: A Randomize Clinical Trial. Iran J Med Sci. 2015 May;40(3):219-24. PMID 25999621
- [Background] Li A, Montano Z, Chen VJ, Gold JI. Virtual reality and pain management: current trends and future directions. Pain Manag. 2011 Mar;1(2):147-157. doi: 10.2217/pmt.10.15. PMID 21779307
- [Background] Treede RD, Rief W, Barke A, Aziz Q, Bennett MI, Benoliel R, Cohen M, Evers S, Finnerup NB, First MB, Giamberardino MA, Kaasa S, Kosek E, Lavand'homme P, Nicholas M, Perrot S, Scholz J, Schug S, Smith BH, Svensson P, Vlaeyen JWS, Wang SJ. A classification of chronic pain for ICD-11. Pain. 2015 Jun;156(6):1003-1007. doi: 10.1097/j.pain.0000000000000160. No abstract available. PMID 25844555
- [Background] Marteau TM, Bekker H. The development of a six-item short-form of the state scale of the Spielberger State-Trait Anxiety Inventory (STAI). Br J Clin Psychol. 1992 Sep;31(3):301-6. doi: 10.1111/j.2044-8260.1992.tb00997.x. PMID 1393159
- [Background] Tashjian VC, Mosadeghi S, Howard AR, Lopez M, Dupuy T, Reid M, Martinez B, Ahmed S, Dailey F, Robbins K, Rosen B, Fuller G, Danovitch I, IsHak W, Spiegel B. Virtual Reality for Management of Pain in Hospitalized Patients: Results of a Controlled Trial. JMIR Ment Health. 2017 Mar 29;4(1):e9. doi: 10.2196/mental.7387. PMID 28356241
- [Background] Mohammed MAA, Khalaf MH, Kesselman A, Wang DS, Kothary N. A Role for Virtual Reality in Planning Endovascular Procedures. J Vasc Interv Radiol. 2018 Jul;29(7):971-974. doi: 10.1016/j.jvir.2018.02.018. PMID 29935787
- [Background] Mosadeghi S, Reid MW, Martinez B, Rosen BT, Spiegel BM. Feasibility of an Immersive Virtual Reality Intervention for Hospitalized Patients: An Observational Cohort Study. JMIR Ment Health. 2016 Jun 27;3(2):e28. doi: 10.2196/mental.5801. PMID 27349654
- [Background] Garrett B, Taverner T, Masinde W, Gromala D, Shaw C, Negraeff M. A rapid evidence assessment of immersive virtual reality as an adjunct therapy in acute pain management in clinical practice. Clin J Pain. 2014 Dec;30(12):1089-98. doi: 10.1097/AJP.0000000000000064. PMID 24535053
- [Background] Tychsen L, Thio LL. Concern of Photosensitive Seizures Evoked by 3D Video Displays or Virtual Reality Headsets in Children: Current Perspective. Eye Brain. 2020 Feb 11;12:45-48. doi: 10.2147/EB.S233195. eCollection 2020. PMID 32104130

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT04687501/Prot_SAP_000.pdf